CLINICAL TRIAL: NCT03376165
Title: Longitudinal Study of Patients Undergoing Cardiac Surgery or Implantation of a Percutaneous Valve Prosthesis
Brief Title: Post-Operative Myocardial Incident & Atrial Fibrillation
Acronym: POMI-AF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: CB2015_75; 2017-A00852-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-11; First posted 2017-12-18 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Valve Heart Disease; Coronary Artery Disease
Keywords: prognosis; translational research
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — for all patients, blood samples with isolation of peripheral blood mononuclear cells, subcutaneous fat
  for patients undergoing cardiac surgery right atrial and left ventricle myocardial samples; Epicardial and mediastinal fat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore predictors of major cardio-vascular events after cardiac surgery and trans-catheter valve implantation with a specific interest in studying mechanisms linking pre-operative leukocyte, fat and myocardial phenotypes with post-intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cardiac surgery (coronary artery bypass graft surgery and/or valvular surgery) or transcatheter valve implantation

Exclusion Criteria:

* pregnant woman
* urgent surgery or intervention
* not able to consent to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients schedulled for cardiac surgery (coronary artery bypass graft surgery and/or valvular surgery) or transcatheter valve implantation and referred to the University Hospital of Lille with inclusion criteria and no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
major cardio-vascular events after cardiac intervention (surgery or transcatheter valve implantation) | from the day of intervention to 10 years
  cardiovascular death, hospitalisation for heart failure, stroke, myocardial infarction, re-intervention

SECONDARY OUTCOMES:
peri-operative myocardial injury | 3 days following intervention
  Area Under the Curve of blood troponin release during the 3 days following cardiac intervention
post-operative myocardial infarction (type 5 myocardial infarction) | 10 days following intervention
  myocardial infarction during the peri-operative time
post-operative atrial fibrillation | 10 days following intervention
  atrial fibrillation onset during post-op hospitalisation
major cardio-vascular events after cardiac intervention (surgery or transcatheter valve implantation) | from the day of intervention to 1 year
  cardiovascular death, hospitalisation for heart failure, stroke, myocardial infarction, re-intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Montaigne, Prof., Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Cardiologie, CHU, Lille, France

REFERENCES:
- [Derived] Ninni S, Vicario R, Coisne A, Woitrain E, Tazibet A, Stewart CM, Diaz LA Jr, White JR, Koussa M, Dubrulle H, Juthier F, Jungling M, Vincentelli A, Edme JL, Nattel S, de Winther M, Geissmann F, Dombrowicz D, Staels B, Montaigne D. Clonal Hematopoiesis Is Associated With Long-Term Adverse Outcomes Following Cardiac Surgery. J Am Heart Assoc. 2024 Sep 3;13(17):e034255. doi: 10.1161/JAHA.123.034255. Epub 2024 Aug 29. PMID 39206728
- [Derived] Ninni S, Dombrowicz D, Kuznetsova T, Vicario R, Gao V, Molendi-Coste O, Haas J, Woitrain E, Coisne A, Neele AE, Prange K, Willemsen L, Aghezzaf S, Fragkogianni S, Tazibet A, Pineau L, White JR, Eeckhoute J, Koussa M, Dubrulle H, Juthier F, Soquet J, Vincentelli A, Edme JL, de Winther M, Geissmann F, Staels B, Montaigne D. Hematopoietic Somatic Mosaicism Is Associated With an Increased Risk of Postoperative Atrial Fibrillation. J Am Coll Cardiol. 2023 Apr 4;81(13):1263-1278. doi: 10.1016/j.jacc.2023.01.036. PMID 36990546